CLINICAL TRIAL: NCT01353274
Title: Survey on Drug Use of Micamlo Combination Tablets AP in Patients With Hypertension
Brief Title: Safety and Efficacy of Daily Use of Micamlo® Combination Tablets AP in Patients With Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1235.38
Record Dates: First submitted 2011-05-09; First posted 2011-05-13 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with hypertension
  Interventions: Drug: Micamlo

INTERVENTIONS:
Drug: Micamlo — Telmisartan plus Amlodipine T40/A5

SUMMARY:
Investigation of safety and efficacy of daily use of Micamlo Combination Tablets AP in patients with Hypertension

ELIGIBILITY:
Inclusion criteria:

- Male and Female patients with hypertension who did not receive of MICAMLO Combination Tablets AP before the start of the study

Exclusion criteria:

* Patients with a history of hypersensitivity to any ingredient of Micamlo Combination Tablets AP and dihydropyridine derivatives
* Pregnant woman or possibly pregnant woman
* Patients with extremely poor bile secretion or patients with serious hepatic disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1200
Sampling Method: Non-Probability Sample
Enrollment: 1157 (Actual)
Dates: Start 2011-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (254):
- Japan (254):
  - Boehringer Ingelheim Investigational Site 199, Akaiwa
  - Boehringer Ingelheim Investigational Site 83, Akishima
  - Boehringer Ingelheim Investigational Site 25, Akita
  - Boehringer Ingelheim Investigational Site 188, Amagasaki
  - Boehringer Ingelheim Investigational Site 116, Anamizu-machi
  - Boehringer Ingelheim Investigational Site 212, Anan
  - Boehringer Ingelheim Investigational Site 145, Anjo
  - Boehringer Ingelheim Investigational Site 11, Aomori
  - Boehringer Ingelheim Investigational Site 12, Aomori
  - Boehringer Ingelheim Investigational Site 192, Arita
  - Boehringer Ingelheim Investigational Site 7, Asahikawa
  - Boehringer Ingelheim Investigational Site 104, Atsugi
  - Boehringer Ingelheim Investigational Site 57, Chiba
  - Boehringer Ingelheim Investigational Site 58, Chiba
  - Boehringer Ingelheim Investigational Site 232, Chikuzen-machi
  - Boehringer Ingelheim Investigational Site 143, Chita
  - Boehringer Ingelheim Investigational Site 23, Daisen
  - Boehringer Ingelheim Investigational Site 24, Daisen
  - Boehringer Ingelheim Investigational Site 10, Date
  - Boehringer Ingelheim Investigational Site 90, Fuchū
  - Boehringer Ingelheim Investigational Site 52, Fujimino
  - Boehringer Ingelheim Investigational Site 129, Fujinomiya
  - Boehringer Ingelheim Investigational Site 103, Fujisawa
  - Boehringer Ingelheim Investigational Site 158, Fukuchiyama
  - Boehringer Ingelheim Investigational Site 224, Fukuoka
  - Boehringer Ingelheim Investigational Site 225, Fukuoka
  - Boehringer Ingelheim Investigational Site 29, Fukushima
  - Boehringer Ingelheim Investigational Site 13, Hachinohe
  - Boehringer Ingelheim Investigational Site 130, Hamamatsu
  - Boehringer Ingelheim Investigational Site 131, Hamamatsu
  - Boehringer Ingelheim Investigational Site 219, Handa
  - Boehringer Ingelheim Investigational Site 171, Hannan
  - Boehringer Ingelheim Investigational Site 204, Hatsukaichi
  - Boehringer Ingelheim Investigational Site 208, Higashihiroshima
  - Boehringer Ingelheim Investigational Site 5, Higashikagura-cho
  - Boehringer Ingelheim Investigational Site 66, Higashimurayama
  - Boehringer Ingelheim Investigational Site 151, Hikone
  - Boehringer Ingelheim Investigational Site 179, Himeji
  - Boehringer Ingelheim Investigational Site 180, Himeji
  - Boehringer Ingelheim Investigational Site 181, Himeji
  - Boehringer Ingelheim Investigational Site 169, Hirakata
  - Boehringer Ingelheim Investigational Site 170, Hirakata
  - Boehringer Ingelheim Investigational Site 201, Hiroshima
  - Boehringer Ingelheim Investigational Site 202, Hiroshima
  - Boehringer Ingelheim Investigational Site 203, Hiroshima
  - Boehringer Ingelheim Investigational Site 38, Hitachi-Naka
  - Boehringer Ingelheim Investigational Site 37, Hitachiota
  - Boehringer Ingelheim Investigational Site 62, Ichikawa
  - Boehringer Ingelheim Investigational Site 17, Ichinoseki
  - Boehringer Ingelheim Investigational Site 223, Iizuka
  - Boehringer Ingelheim Investigational Site 175, Ikeda
  - Boehringer Ingelheim Investigational Site 238, Iki
  - Boehringer Ingelheim Investigational Site 63, IKisarazu
  - Boehringer Ingelheim Investigational Site 191, Ikoma
  - Boehringer Ingelheim Investigational Site 111, Imizu
  - Boehringer Ingelheim Investigational Site 189, Itami
  - Boehringer Ingelheim Investigational Site 253, Itoman
  - Boehringer Ingelheim Investigational Site 233, Itoshima
  - Boehringer Ingelheim Investigational Site 252, Izumi
  - Boehringer Ingelheim Investigational Site 249, Kagoshima
  - Boehringer Ingelheim Investigational Site 250, Kagoshima
  - Boehringer Ingelheim Investigational Site 125, Kakamigahara
  - Boehringer Ingelheim Investigational Site 229, Kama
  - Boehringer Ingelheim Investigational Site 152, Kameoka
  - Boehringer Ingelheim Investigational Site 241, Kamiamakusa
  - Boehringer Ingelheim Investigational Site 242, Kamiamakusa
  - Boehringer Ingelheim Investigational Site 22, Kamimachi
  - Boehringer Ingelheim Investigational Site 113, Kanazawa
  - Boehringer Ingelheim Investigational Site 114, Kanazawa
  - Boehringer Ingelheim Investigational Site 237, Kanzaki
  - Boehringer Ingelheim Investigational Site 144, Kariya
  - Boehringer Ingelheim Investigational Site 33, Kasama
  - Boehringer Ingelheim Investigational Site 34, Kasama
  - Boehringer Ingelheim Investigational Site 137, Kasugai
  - Boehringer Ingelheim Investigational Site 138, Kasugai
  - Boehringer Ingelheim Investigational Site 48, Kasukabe
  - Boehringer Ingelheim Investigational Site 49, Kasukabe
  - Boehringer Ingelheim Investigational Site 177, Katō
  - Boehringer Ingelheim Investigational Site 178, Katō
  - Boehringer Ingelheim Investigational Site 117, Katsuyama
  - Boehringer Ingelheim Investigational Site 121, Kawachi-Nagano
  - Boehringer Ingelheim Investigational Site 51, Kawaguchi
  - Boehringer Ingelheim Investigational Site 100, Kawasaki
  - Boehringer Ingelheim Investigational Site 101, Kawasaki
  - Boehringer Ingelheim Investigational Site 43, Kiryū
  - Boehringer Ingelheim Investigational Site 176, Kita-ku
  - Boehringer Ingelheim Investigational Site 15, Kitakami
  - Boehringer Ingelheim Investigational Site 226, Kitakyushu
  - Boehringer Ingelheim Investigational Site 227, Kitakyushu
  - Boehringer Ingelheim Investigational Site 4, Kitami
  - Boehringer Ingelheim Investigational Site 183, Kobe
  - Boehringer Ingelheim Investigational Site 184, Kobe
  - Boehringer Ingelheim Investigational Site 185, Kobe
  - Boehringer Ingelheim Investigational Site 186, Kobe
  - Boehringer Ingelheim Investigational Site 187, Kobe
  - Boehringer Ingelheim Investigational Site 220, Kochi
  - Boehringer Ingelheim Investigational Site 56, Koshigaya
  - Boehringer Ingelheim Investigational Site 193, Kotoura-cho
  - Boehringer Ingelheim Investigational Site 240, Kotouracho
  - Boehringer Ingelheim Investigational Site 30, Kōriyama
  - Boehringer Ingelheim Investigational Site 53, Kumagaya
  - Boehringer Ingelheim Investigational Site 243, Kumamoto
  - Boehringer Ingelheim Investigational Site 196, Kurashiki
  - Boehringer Ingelheim Investigational Site 205, Kure
  - Boehringer Ingelheim Investigational Site 206, Kure
  - Boehringer Ingelheim Investigational Site 230, Kurume
  - Boehringer Ingelheim Investigational Site 231, Kurume
  - Boehringer Ingelheim Investigational Site 149, Kusatsu
  - Boehringer Ingelheim Investigational Site 9, Kushiro
  - Boehringer Ingelheim Investigational Site 153, Kyoto
  - Boehringer Ingelheim Investigational Site 154, Kyoto
  - Boehringer Ingelheim Investigational Site 155, Kyoto
  - Boehringer Ingelheim Investigational Site 156, Kyoto
  - Boehringer Ingelheim Investigational Site 157, Kyoto
  - Boehringer Ingelheim Investigational Site 99, Matsuda-machi
  - Boehringer Ingelheim Investigational Site 64, Matsudo
  - Boehringer Ingelheim Investigational Site 65, Matsudo
  - Boehringer Ingelheim Investigational Site 195, Matsue
  - Boehringer Ingelheim Investigational Site 119, Matsumoto
  - Boehringer Ingelheim Investigational Site 120, Matsumoto
  - Boehringer Ingelheim Investigational Site 234, Matsuura
  - Boehringer Ingelheim Investigational Site 216, Matsuyama
  - Boehringer Ingelheim Investigational Site 217, Matsuyama
  - Boehringer Ingelheim Investigational Site 148, Matsuzaka
  - Boehringer Ingelheim Investigational Site 207, Mihara
  - Boehringer Ingelheim Investigational Site 122, Minamiminowa-mura
  - Boehringer Ingelheim Investigational Site 248, Miyazaki
  - Boehringer Ingelheim Investigational Site 126, Mizunami
  - Boehringer Ingelheim Investigational Site 60, Mobara
  - Boehringer Ingelheim Investigational Site 61, Mobara
  - Boehringer Ingelheim Investigational Site 16, Morioka
  - Boehringer Ingelheim Investigational Site 27, Murayama
  - Boehringer Ingelheim Investigational Site 105, Nagaoka
  - Boehringer Ingelheim Investigational Site 106, Nagaoka
  - Boehringer Ingelheim Investigational Site 235, Nagasaki
  - Boehringer Ingelheim Investigational Site 254, Nago
  - Boehringer Ingelheim Investigational Site 139, Nagoya
  - Boehringer Ingelheim Investigational Site 140, Nagoya
  - Boehringer Ingelheim Investigational Site 141, Nagoya
  - Boehringer Ingelheim Investigational Site 142, Nagoya
  - Boehringer Ingelheim Investigational Site 228, Nakagawamachi
  - Boehringer Ingelheim Investigational Site 39, Nakagawamachi
  - Boehringer Ingelheim Investigational Site 245, Nakatsu
  - Boehringer Ingelheim Investigational Site 127, Nakatsugawa
  - Boehringer Ingelheim Investigational Site 59, Narita
  - Boehringer Ingelheim Investigational Site 18, Natori
  - Boehringer Ingelheim Investigational Site 8, Nayoro
  - Boehringer Ingelheim Investigational Site 246, Nichinan
  - Boehringer Ingelheim Investigational Site 31, Nihonmatsu
  - Boehringer Ingelheim Investigational Site 107, Niigata
  - Boehringer Ingelheim Investigational Site 200, Niimi
  - Boehringer Ingelheim Investigational Site 6, Nikki-cho
  - Boehringer Ingelheim Investigational Site 128, Nishiizu-cho
  - Boehringer Ingelheim Investigational Site 182, Nishinomiya
  - Boehringer Ingelheim Investigational Site 112, Nomi
  - Boehringer Ingelheim Investigational Site 134, Numazu
  - Boehringer Ingelheim Investigational Site 197, Okayama
  - Boehringer Ingelheim Investigational Site 198, Okayama
  - Boehringer Ingelheim Investigational Site 14, Omamachi
  - Boehringer Ingelheim Investigational Site 159, Osaka
  - Boehringer Ingelheim Investigational Site 160, Osaka
  - Boehringer Ingelheim Investigational Site 161, Osaka
  - Boehringer Ingelheim Investigational Site 162, Osaka
  - Boehringer Ingelheim Investigational Site 163, Osaka
  - Boehringer Ingelheim Investigational Site 164, Osaka
  - Boehringer Ingelheim Investigational Site 165, Osaka
  - Boehringer Ingelheim Investigational Site 166, Osaka
  - Boehringer Ingelheim Investigational Site 167, Osaka
  - Boehringer Ingelheim Investigational Site 168, Osaka
  - Boehringer Ingelheim Investigational Site 40, Oyama
  - Boehringer Ingelheim Investigational Site 26, Ōdate
  - Boehringer Ingelheim Investigational Site 124, Ōgaki
  - Boehringer Ingelheim Investigational Site 244, Ōita
  - Boehringer Ingelheim Investigational Site 239, Ōmura
  - Boehringer Ingelheim Investigational Site 35, Ryūgasaki
  - Boehringer Ingelheim Investigational Site 236, Saga
  - Boehringer Ingelheim Investigational Site 102, Sagamihara
  - Boehringer Ingelheim Investigational Site 46, Saitama
  - Boehringer Ingelheim Investigational Site 47, Saitama
  - Boehringer Ingelheim Investigational Site 172, Sakai
  - Boehringer Ingelheim Investigational Site 173, Sakai
  - Boehringer Ingelheim Investigational Site 215, Sakaidechō
  - Boehringer Ingelheim Investigational Site 118, Sakakimachi
  - Boehringer Ingelheim Investigational Site 108, Sanjyo
  - Boehringer Ingelheim Investigational Site 41, Sano
  - Boehringer Ingelheim Investigational Site 1, Sapporo
  - Boehringer Ingelheim Investigational Site 2, Sapporo
  - Boehringer Ingelheim Investigational Site 3, Sapporo
  - Boehringer Ingelheim Investigational Site 55, Sayama
  - Boehringer Ingelheim Investigational Site 21, Sendai
  - Boehringer Ingelheim Investigational Site 115, Shikamachichō-shimoutagaura
  - Boehringer Ingelheim Investigational Site 210, Shimonoseki
  - Boehringer Ingelheim Investigational Site 19, Shiogama
  - Boehringer Ingelheim Investigational Site 32, Shirakawa
  - Boehringer Ingelheim Investigational Site 132, Shizuoka
  - Boehringer Ingelheim Investigational Site 133, Shizuoka
  - Boehringer Ingelheim Investigational Site 50, Sōka
  - Boehringer Ingelheim Investigational Site 174, Suita
  - Boehringer Ingelheim Investigational Site 147, Suzuka
  - Boehringer Ingelheim Investigational Site 69, Tachikawa
  - Boehringer Ingelheim Investigational Site 70, Tachikawa
  - Boehringer Ingelheim Investigational Site 71, Tachikawa
  - Boehringer Ingelheim Investigational Site 20, Tagajyo
  - Boehringer Ingelheim Investigational Site 44, Takasaki
  - Boehringer Ingelheim Investigational Site 45, Takasaki
  - Boehringer Ingelheim Investigational Site 150, Takashima
  - Boehringer Ingelheim Investigational Site 84, Tama
  - Boehringer Ingelheim Investigational Site 28, Tendō
  - Boehringer Ingelheim Investigational Site 213, Tokushima
  - Boehringer Ingelheim Investigational Site 72, Tokyo Adachi-ku
  - Boehringer Ingelheim Investigational Site 73, Tokyo Adachi-ku
  - Boehringer Ingelheim Investigational Site 74, Tokyo Bunkyo-ku
  - Boehringer Ingelheim Investigational Site 75, Tokyo Bunkyo-ku
  - Boehringer Ingelheim Investigational Site 79, Tokyo Chuo-ku
  - Boehringer Ingelheim Investigational Site 77, Tokyo Edofawa-ku
  - Boehringer Ingelheim Investigational Site 76, Tokyo Itabashi-ku
  - Boehringer Ingelheim Investigational Site 89, Tokyo Katsushika-ku
  - Boehringer Ingelheim Investigational Site 85, Tokyo Meguro-ku
  - Boehringer Ingelheim Investigational Site 86, Tokyo Meguro-ku
  - Boehringer Ingelheim Investigational Site 81, Tokyo Nerima-ku
  - Boehringer Ingelheim Investigational Site 82, Tokyo Nerima-ku
  - Boehringer Ingelheim Investigational Site 87, Tokyo Ota-ku
  - Boehringer Ingelheim Investigational Site 67, Tokyo Shinjyuku-ku
  - Boehringer Ingelheim Investigational Site 68, Tokyo Shinjyuku-ku
  - Boehringer Ingelheim Investigational Site 78, Tokyo Sumida-ku
  - Boehringer Ingelheim Investigational Site 88, Tokyo Sumida-ku
  - Boehringer Ingelheim Investigational Site 80, Tokyo Toshima-ku
  - Boehringer Ingelheim Investigational Site 214, Tonosho-cho
  - Boehringer Ingelheim Investigational Site 221, Tosashimizu
  - Boehringer Ingelheim Investigational Site 110, Toyama
  - Boehringer Ingelheim Investigational Site 135, Toyohashi
  - Boehringer Ingelheim Investigational Site 136, Toyohashi
  - Boehringer Ingelheim Investigational Site 109, Tōkamachi
  - Boehringer Ingelheim Investigational Site 146, Tsu
  - Boehringer Ingelheim Investigational Site 36, Tsuchiura
  - Boehringer Ingelheim Investigational Site 247, Tsunocho
  - Boehringer Ingelheim Investigational Site 209, Ube
  - Boehringer Ingelheim Investigational Site 123, Ueda
  - Boehringer Ingelheim Investigational Site 42, Utsunomiya
  - Boehringer Ingelheim Investigational Site 218, Uwajima
  - Boehringer Ingelheim Investigational Site 251, Wadomari
  - Boehringer Ingelheim Investigational Site 211, Yamaguchi
  - Boehringer Ingelheim Investigational Site 190, Yamatokooriyama
  - Boehringer Ingelheim Investigational Site 222, Yame
  - Boehringer Ingelheim Investigational Site 93, Yokohama
  - Boehringer Ingelheim Investigational Site 94, Yokohama
  - Boehringer Ingelheim Investigational Site 95, Yokohama
  - Boehringer Ingelheim Investigational Site 96, Yokohama
  - Boehringer Ingelheim Investigational Site 97, Yokohama
  - Boehringer Ingelheim Investigational Site 91, Yokosuka
  - Boehringer Ingelheim Investigational Site 92, Yokosuka
  - Boehringer Ingelheim Investigational Site 54, Yokoze-machi
  - Boehringer Ingelheim Investigational Site 194, Yonago
  - Boehringer Ingelheim Investigational Site 98, Zama

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Hypertension: Micamlo Combination Tablets AP: Telmisartan 40 mg plus Amlodipine 5 mg, oral administration
Period: Overall Study
Arm/Group | Patients With Hypertension
Started | 1157
Completed | 1129
Not Completed | 28
Not completed — No case report form (CRF) collected | 28

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Hypertension
Number analyzed (Participants) | 1109
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 514
  Male | 595

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Drug-related Adverse Events
Description: Number of patients with drug-related adverse events
Time Frame: 12 months
Population: Safety set: all patients who were documented to have taken at least one dose of T40/A5 mg FDC except for patients who had no observation documented after entry, made invalid registration or were not under the appropriate site contact
Measure: Number; unit: participants
Arm/Group | Patients With Hypertension
Number analyzed (Participants) | 1109
participants | 60

2. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP)
Description: Change from baseline in SBP after 1, 2, 3, 6, 12 months
Time Frame: after 1, 2, 3, 6, 12 months
Population: Efficacy set: all patients in the safety set who were labelled by T40/A5 mg Fixed Dose Combination (FDC) and have analysable BP data at baseline and at least one post-baseline time point. Missing data were imputed using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients With Hypertension
Number analyzed (Participants) | 1108
mmHg
  Month 1 | -15.9 (18.5)
  Month 2 | -16.5 (18.6)
  Month 3 | -16.7 (19.5)
  Month 6 | -17.7 (20.0)
  Month 12 | -19.2 (19.7)

3. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP)
Description: Change from baseline in DBP after 1, 2, 3, 6, 12 months
Time Frame: after 1, 2, 3, 6, 12 months
Population: Efficacy set: all patients in the safety set who were labelled by T40/A5 mg FDC and have analysable BP data at baseline and at least one post-baseline time point. Missing data were imputed using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients With Hypertension
Number analyzed (Participants) | 1108
mmHg
  Month 1 | -7.6 (11.7)
  Month 2 | -8.4 (12.2)
  Month 3 | -8.2 (12.2)
  Month 6 | -8.9 (12.7)
  Month 12 | -9.8 (12.5)

4. Secondary Outcome: Proportion of Patients Who Achieved the Target BP
Description: Proportion of patients who achieved the target BP after 1, 2, 3, 6, 12 months
Time Frame: after 1, 2, 3, 6, 12 months
Population: as for outcome 3
Measure: Number; unit: Percentage of patients (target BP)
Arm/Group | Patients With Hypertension
Number analyzed (Participants) | 1108
Percentage of patients (target BP)
  Month 1 | 54.2
  Month 2 | 57.8
  Month 3 | 58.8
  Month 6 | 62.4
  Month 12 | 66.5

5. Secondary Outcome: Proportion of Patients Who Normalised Their BP
Description: Proportion of patients who normalised their BP after 1, 2, 3, 6, 12 months
Time Frame: after 1, 2, 3, 6, 12 months
Population: as for outcome 3
Measure: Number; unit: Percentage of patients (normalised BP)
Arm/Group | Patients With Hypertension
Number analyzed (Participants) | 1108
Percentage of patients (normalised BP)
  Month 1 | 61.3
  Month 2 | 66.3
  Month 3 | 67.2
  Month 6 | 70.4
  Month 12 | 73.7

ADVERSE EVENTS:
Time Frame: During the 12-month period under the administration of T40/A5 mg FDC, up to 95 weeks
Arm/Group | Patients With Hypertension
Serious Adverse Events (participants affected / at risk) | 22/1109
Other Adverse Events (participants affected / at risk) | 0/1109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Hypertension (N=1109)
Acute myocardial infarction (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrage (Gastrointestinal disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Nephrosclerosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Aortic dissection (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.